CLINICAL TRIAL: NCT02682264
Title: An Open-Label, Long-Term Extension Study to Evaluate the Safety of Cortexolone 17α-Propionate (CB-03-01) Cream, 1% Applied Twice-Daily in Subjects With Acne Vulgaris
Brief Title: An Open-Label, Long-Term Extension Study to Evaluate the Safety of CB-03-01 Cream, 1% in Participants With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cassiopea SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-03-01/27
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Acne Vulgaris
Keywords: acne; clascoterone; anti-androgen
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CB-03-01 cream, 1% (Experimental): CB-03-01 (cortexolone 17α-propionate) Cream, 1%, applied twice daily to whole face (about 1 gram) and affected areas of trunk (if applicable) for up to an additional 9 months. Over the course of the study, treatment on the face and/or trunk may be discontinued if/when acne clears and re-started if/when acne worsens, according to the assessment of the investigator for each respective treatment area.
  Interventions: Drug: CB-03-01 cream, 1%

INTERVENTIONS:
Drug: CB-03-01 cream, 1% — Cortexolone 17α-propionate (USAN/INN: clascoterone) is a steroidal antiandrogen that is being developed as a 1% cream for the topical treatment of acne vulgaris.
  Other Names: cortexolone 17α-propionate; clascoterone (USAN, INN)

SUMMARY:
The primary objective of this study is to determine the long-term safety of CB-03-01 cream, 1% applied twice daily for an additional nine months in study participants with acne vulgaris that participated in the Phase 3 pivotal studies for a total treatment of up to 12 months.

DETAILED DESCRIPTION:
This was a multicenter, open label, long-term extension study for CB-03-01 cream, 1% focused on safety in male and female participants, 9 years or older who completed one of the Phase 3 pivotal studies [CB-03-01/25 and CB-03-01/26]. Participants applies the active medication (CB-03-01 cream, 1%) twice daily to the entire face and, if designated by investigator AND desired by the participant, truncal acne for nine additional months of treatment. Thus, overall participants were exposed to CB-03-01 cream, 1% for a total treatment of up to 12 months (0 or 3 months in the Phase 3 pivotal study and an additional nine months in this long-term safety study).

Participants treated facial acne per protocol for nine months. Treatment of truncal acne was discussed by the investigator and participant. Treatment on the face and/or trunk was discontinued if/when acne clears and re-started if/when acne worsens, according to the assessment of the investigator for each respective treatment area (i.e., face and trunk).

Participants were rolled over from the Phase 3 pivotal studies [CB-03-01/25 and CB-03-01/26] into this long-term, safety study in order to achieve at least 300 participants on-study at 6 months and 100 participants on-study at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant has successfully completed participation in one of the Phase 3 pivotal studies [CB-03-01/25 and CB-03-01/26].
* Participant agrees to use effective method of contraception throughout study, if applicable.
* Participant has provided written informed consent or assent.
* Participant is willing to comply with study instructions and return to the clinic for required visits.

Exclusion Criteria:

* Participant is pregnant, lactating, or is planning to become pregnant during the study.
* Participant has any skin disease or condition that could interfere with the safety evaluation of the test products or requires the use of interfering topical or systemic therapy.
* Participant has any condition which, in the investigator's opinion, would make it unsafe or unsuitable for the participant to participate in this research study.
* Participant plans to use any other investigational drug or device during participation in this study.
* Participant has known hypersensitivity or previous allergic reaction to the drug or any of its ingredients.
* Participant is or plans to use any restricted systemic and/or topical anti-acne preparations or medications during the study

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R&D Cassiopea, Study Director — Cassiopea SpA
Locations (74):
- United States (39):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Gary M. Petrus, MD PA, Little Rock, Arkansas
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Rady Childrens Hospital, Pediatric and Adolescent Dermatology, San Diego, California
  - Southern California Dermatology, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Memorial Research Medical Clinic dba / Orange County Research Center, Tustin, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Study Protocol, Inc., Boynton Beach, Florida
  - Tory Sullivan, M.D., P.A., North Miami Beach, Florida
  - Belleair Research Center, Pinellas Park, Florida
  - Meridien Research, St. Petersburg, Florida
  - MOORE Clinical Research, Inc., Tampa, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Arlington Dermatology, Arlington Heights, Illinois
  - Shideler Clinical Research Center, Carmel, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Maryland Laser Skin and Vein Institute, Hunt Valley, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Sadick Research Group, LLC, New York, New York
  - Skin Specialty Dermatology, New York, New York
  - DermResearch Center of New York, Inc., Stony Brook, New York
  - Oregon Dermatology and Research Center, Portland, Oregon
  - The Pennsylvania State University and the Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Greenville Dermatology, LLC, Greenville, South Carolina
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Westlake Dermatology Clinical Research Center, Austin, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Clinical Research Associates of Tidewater, Inc., Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
- Bulgaria (6):
  - Site 3521, Plovdiv
  - 3520, Sofia
  - Site 3524, Sofia
  - Site 3519, Sofia
  - Site 3526, Sofia
  - Site 3522, Varna
- Georgia (3):
  - Site 9912, Tbilisi
  - Site 9911, Tbilisi
  - Site 9913, Tbilisi
- Poland (11):
  - Site 4814, Bialystok
  - 4819, Bydgoszcz
  - Site 4822, Częstochowa
  - Site 4811, Dąbrówka
  - 4815, Katowice
  - Site 4821, Krakow
  - Site 4820, Lodz
  - Site 4823, Osielsko
  - Site 4813, Szczecin
  - Site 4818, Warsaw
  - Site 4812, Wroclaw
- Romania (8):
  - Site 4033, Sector 2, Bucharest
  - Site 4034, Sector 2, Bucharest
  - Site 4031, Sector 3, Bucharest
  - Site 4029, Sector 6, Bucharest
  - Site 4028, Târgovişte, Jud. Dambovita
  - Site 4035, Bucharest
  - Site 4037, Iași
  - Site 4030, Sibiu
- Serbia (3):
  - Site 8138, Belgrade
  - Site 8137, Belgrade
  - Site 8136, Novi Sad
- Ukraine (4):
  - Site 3802, Dnipro
  - Site 3808, Kharkiv
  - Site 3804, Kharkiv
  - Site 3809, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 609 subjects who were rolled over (i.e., enrolled) from the two Phase 3 pivotal studies (CB-03-01/25 [NCT02608450] and CB-03-01/26 [NCT02608476]) into this long-term, safety study. However, two (2) subjects in the original vehicle cream were not treated with test article and thus were excluded from the study population (Safety set).
Groups:
- CB-03-01 Cream, 1%: Subjects in this arm received CB-03-01 (cortexolone 17α-propionate) Cream, 1% in the pivotal study and continued their CB-03-01 cream treatment in this open-label safety extension study. Subjects were instructed to apply CB-03-01 Cream, 1%, twice daily to whole face (about 1 gram) and affected areas of trunk (if applicable) for up to an additional 9 months. Over the course of the study, treatment on the face and/or trunk may be discontinued if/when acne clears and re-started if/when acne worsens, according to the assessment of the investigator for each respective treatment area.
  Cortexolone 17α-propionate (USAN/INN: clascoterone) is a steroidal antiandrogen that is being developed as a 1% cream for the topical treatment of acne vulgaris.
- CB-03-01 Cream, 1% (Vehicle Arm): Subjects in this arm received vehicle cream in the pivotal study and CB-03-01 cream in this open-label safety extension study.
Period: Overall Study
Arm/Group | CB-03-01 Cream, 1% | CB-03-01 Cream, 1% (Vehicle Arm)
Started | 317 | 290
Completed | 179 | 168
Not Completed | 138 | 122
Not completed — Withdrawal by Subject | 56 | 45
Not completed — Lost to Follow-up | 49 | 41
Not completed — Lack of Efficacy | 14 | 16
Not completed — Withdrawal by Parent | 6 | 7
Not completed — Adverse Event | 9 | 0
Not completed — Noncompliance with study drug | 1 | 4
Not completed — Pregnancy | 1 | 2
Not completed — Recovery | 1 | 2
Not completed — Progressive Disease | 1 | 0
Not completed — Technical Problems | 0 | 1
Not completed — Moved abroad and unable to continue | 0 | 3
Not completed — Stopped test article application | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population defined as all subjects who applied at least one dose of test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | CB-03-01 Cream, 1% | CB-03-01 Cream, 1% (Vehicle Arm) | Total
Number analyzed (Participants) | 317 | 290 | 607
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.2 (5.8) | 19.3 (6.7) | 19.2 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 183 | 381
  Male | 119 | 107 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 15 | 42
  Not Hispanic or Latino | 290 | 275 | 565
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 8 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 17 | 18 | 35
  White | 283 | 256 | 539
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Local and Systemic Treatment Emergent Adverse Events
Description: Number of participants with any local and systemic treatment emergent AEs (TEAEs)
Time Frame: up to 52 weeks
Population: Safety dataset population.
Measure: Count of Participants; unit: Participants
Arm/Group | CB-03-01 Cream, 1% | CB-03-01 Cream, 1% (Vehicle Arm)
Number analyzed (Participants) | 317 | 290
Participants | 58 | 52

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) were collected from the time the subject exited the pivotal study (i.e., Week 13 or day 1 of the Long-term extension study) and up to 52 weeks after entry into the pivotal study (i.e., up to week 39 or early termination of the long term extension study).
Arm/Group | CB-03-01 Cream, 1% | CB-03-01 Cream, 1% (Vehicle Arm)
All-Cause Mortality (participants affected / at risk) | 0/317 | 0/290
Serious Adverse Events (participants affected / at risk) | 3/317 | 3/290
Other Adverse Events (participants affected / at risk) | 21/317 | 17/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-03-01 Cream, 1% (N=317) | CB-03-01 Cream, 1% (Vehicle Arm) (N=290)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery dissection (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-03-01 Cream, 1% (N=317) | CB-03-01 Cream, 1% (Vehicle Arm) (N=290)
Nasopharyngitis (Infections and infestations) | 6 (7) | 10 (13)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 4 (4)
Sinusitis (Infections and infestations) | 3 (3) | 2 (2)
Application site acne (General disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 18 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 60 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-09-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02682264/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT02682264/SAP_001.pdf